CLINICAL TRIAL: NCT02640326
Title: A Prospective Randomized Control Trial Comparing Routine Urinary Catheterization vs. No-Urinary Catheterization at the Time of Thoracoscopic Pulmonary Resection (McMaster Catheterization for Thoracoscopic Surgery Study - UCATh Study)
Brief Title: McMaster Catheterization for Thoracoscopic Surgery Study
Acronym: UCATh
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Research question no longer useful/feasible due to shifts in standards of care
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SJHH_UCATh
Record Dates: First submitted 2015-12-22; First posted 2015-12-28 (Estimated); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Non-Small Cell Lung Cancer; Lung Neoplasms; Metastatic Lung Cancer; Urinary Retention; Urinary Tract Infections
Keywords: Urinary Catheterization; Randomized Controlled Trial; Thoracic Surgery, Video-Assisted; Quality Improvement; Evidence-Based Practice; Post-operative complications
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Urinary Retention; Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator (Active Comparator): The catheterized arm will have Standard of care Foley urinary catheter insertion according to usual institutional care pathways in the operating room prior to surgery initiation. The urinary catheter will be assessed for removal on the morning of post-operative day 1, and patients will be monitored for urinary complications once catheter is removed until patient has successfully voided spontaneously within 8 +/- 2 hours.
  Interventions: Other: No Foley Urinary Catheter
- Experimental Arm (Experimental): The non-catheterized arm will have standard of care Foley urinary catheter insertion, with no Foley Urinary Catheter inserted prior to, during, or after surgery unless the patient is showing signs of urinary retention after surgery. Patient will be monitored for urinary complications starting in the recovery room until patient has successfully voided spontaneously within 8 +/- 2 hours
  Interventions: Other: Standard of care Foley urinary catheter insertion

INTERVENTIONS:
Other: No Foley Urinary Catheter — No Foley urinary catheter will be put in place during the operation
  Other Names: Experimental Comparator
  Arms: Active Comparator
Other: Standard of care Foley urinary catheter insertion — A Foley urinary catheter will be put in place during the operation
  Other Names: Active Comparator
  Arms: Experimental Arm

SUMMARY:
It is common practice to insert a Foley catheter into the bladder to drain urine during and after a lung resection. Recently, there has been increasing interest in the potential risks associated with this catheterization, particularly with regard to infection. As thoracic surgery adopts minimally invasive surgical techniques, the need for urinary catheterization during surgery is being questioned since these less invasive surgeries are known to result in less post-operative acute pain, shorter length of stay, and other outcomes that tend to decrease overall anesthetic needs for this patient population. Thus, there is a need to investigate whether patients who have had a minimally invasive lung resection truly need the Foley catheter at all. This will be achieved by assigning patients to either an experimental no-catheter group or the standard of care routine urinary catheter group to determine if patients with no catheter experience different rates of complications. This pilot study will primarily determine if there is a difference in post operative urinary complications between the groups. It is hoped that this study will definitively determine whether a Foley urine catheter is a necessary procedure in the course of a minimally invasive lung resection.

DETAILED DESCRIPTION:
Urinary catheterization is standard practice during and shortly after lung resections. The standard practice is being questioned in an era where unnecessary interventions are being re-considered, particularly since urinary catheterization is not without a risk of adverse events. The study is being done to establish an evidence base to support widespread discontinuation or continuation of this standard practice. Consenting patients will be randomized to either the catheterized or non-catheterized arms. Patient urinary management will be managed as per an a priori-defined protocol that follows St. Joseph's Healthcare Hamilton (SJHH) institutional standards.

ELIGIBILITY:
Inclusion Criteria:

* Must undergo minimally invasive Video-Assisted Thoracoscopic Thoracic Surgery (VATS) or Robotic-Assisted Thoracoscopic Thoracic Surgery (RTS) anatomic pulmonary resection surgery (lobectomy, segmentectomy)
* Must be diagnosed with primary or secondary lung cancer eligible for resection

Exclusion Criteria:

* Patients who are unwilling to comply with study procedures
* Patients who are unable to complete questionnaires with assistance
* Non-VATS/RTS pulmonary resection patients
* Non-anatomic pulmonary resection
* Patients with benign disease
* Patients requiring chronic urinary catheterization
* Patients with contraindications to placement of urinary catheter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Postoperative urinary complications | From the time of surgery to post-operative Day 14.
  Compating the difference in the rate of the occurrence of one or more of postoperative urinary tract infection, postoperative urinary retention requiring 1 catheterization, and postoperative urinary retention requiring more than 1 catheterization between the catheterized and the non-catheterized arms

SECONDARY OUTCOMES:
Length of Hospital Stay | During patient hospital stay (Estimated to be between post-operative day 0 and day 7)
  Comparing the total length of hospital stay between the catheterized and non-catheterized arms
Rate of Post-operative Hypotension | During patient hospital stay (Estimated to be between post-operative day 0 and day 7)
  Post-operative hypotension will be defined as systolic blood pressure less than 80 mmHg for > 6 hours requiring active fluid resuscitation. The comparison will be made of rate of occurrence between the catheterized and non-catheterized arms to account for varied volumes of fluid intake that may confound observations
Total IV fluid administration | First 48 hours of the perioperative period
  The comparison will be made of rate of occurrence between the catheterized and non-catheterized arms to account for varied volumes of fluid intake that may confound observations
Validity of the bladder scanner tool relative to actual urine output | During patient hospital stay (Estimated to be between post-operative day 0 and day 7)
  In patients who underwent a bladder scan for suspected urinary retention (Failure to pass urine within 8 +/-2 hours of de-catheterization or after surgery), it is necessary to measure how accurate the bladder scan procedure is relative to the actual amount of urine in the bladder. The bladder scanner will generate an estimate of the amount of urine in the bladder, but the accuracy is not known. The volume of urine collected from the catheter by nursing staff or as measured from a urine collection hat and compared to the reading from the bladder scanner
Rate of peri-operative pulmonary complications | During patient hospital stay (Estimated to be between post-operative day 0 and day 7)
  Pulmonary complications defined as Grade II or greater according to the Ottawa Thoracic Morbidity and Mortality (TM&M) scale (requiring treatment). The comparison will be made of rate of complication occurrence between the catheterized and non-catheterized arms
Rate of peri-operative cardiac complications | During patient hospital stay (Estimated to be between post-operative day 0 and day 7)
  Cardiac complications defined as Grade I or greater according to the Ottawa Thoracic Morbidity and Mortality (TM&M) scale (no treatment required). The comparison will be made of rate of complication occurrence between the catheterized and non-catheterized arms

CONTACTS AND LOCATIONS:
Overall Officials: John Agzarian, MD, MPH, FRCSC, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No